CLINICAL TRIAL: NCT04339062
Title: Safety and Efficacy of Cemiplimab (PD-1 Blockade) in Selected Organ Transplant Recipients With Advanced Cutaneous Squamous Cell Carcinoma (CONTRAC)
Brief Title: Cemiplimab in AlloSCT/SOT Recipients With CSCC
Acronym: CONTRAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-817
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Advanced Cancer
Keywords: Cutaneous Squamous Cell Carcinoma; Advanced Cancer; Allogeneic hematopoietic stem cell transplant; Kidney transplant
MeSH Terms: interventions — cemiplimab; Everolimus; Sirolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 Cemiplimab (Experimental): Participants who received allogeneic hematopoietic stem cell transplant
  -- Cemiplimab: via IV, flat predetermined dosage every 21 days
  Interventions: Drug: Cemiplimab
- Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone (Experimental): Participants who received a kidney transplant will receive
  * Cemiplimab via IV, flat predetermined dosage every 21 days
  * Everolimus or Sirolimus-least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  * Prednisone 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapering doses while receiving Cemiplimab
  Interventions: Drug: Cemiplimab; Drug: Everolimus; Drug: Sirolimus; Drug: Prednisone

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab: via IV, flat predetermined dosage every 21 days.
  Other Names: Libtayo
Drug: Everolimus — Everolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Other Names: Afinitor; Zortress
  Arms: Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Drug: Sirolimus — Sirolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Other Names: Rapamune
  Arms: Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Drug: Prednisone — 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapered dosing while receiving Cemiplimab
  Other Names: Deltasone; Prednicot; predniSONE Intensol; Rayos; Sterapred; Sterapred DS
  Arms: Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone

SUMMARY:
In this research study, Cemiplimab is being evaluated as a treatment for advanced cutaneous squamous cell carcinoma in participants who have previously received an allogeneic hematopoietic stem cell transplant or kidney transplant.

- This research study involves the following drug(s):

* Cemiplimab
* Everolimus or Sirolimus
* Prednisone

DETAILED DESCRIPTION:
* This an open-label, two cohort, phase I/II research study to evaluate the safety and effectiveness of Cemiplimab as a treatment for advanced cutaneous squamous cell carcinoma in participants who have received allogeneic hematopoietic stem cell or kidney transplants.
* The research study procedures include screening for eligibility, study treatment, participant evaluations and safety follow-up visits. It is expected that about 12 people will take part in this research study.

  * Participants will be divided into two groups (cohorts) of allogeneic hematopoietic stem cell recipients or kidney transplants recipients.
  * Allogeneic hematopoietic stem cell recipients will only receive the study treatment drug of Cemiplimab.
  * Kidney transplant recipients will receive the study treatment drug of Cemiplimab along with the immunosuppressant drugs of Everolimus or Sirolimus and Prednisone to prevent kidney rejection.

The U.S. Food and Drug Administration (FDA) has approved Cemiplimab as a treatment option for patients with advanced cutaneous squamous cell cancer, but the FDA has not approved the use of Cemiplimab in participants who have received allogeneic hematopoietic stem cell transplants or kidney transplants in the past.

-- Cemiplimab is a type of drug called a monoclonal antibody. Antibodies are proteins naturally found in your blood that fight infections. A monoclonal antibody is a special kind of antibody that is manufactured as a medication to target specific proteins in the body that may be involved this type of cancer.

Cemiplimab is a human monoclonal anti-PD-1 antibody that works by blocking the programmed death-1 (PD-1), a cell receptor on immune cells that is involved in preventing immune cells from destroying other cells. Blocking the receptor is expected to help immune cells attack cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, advanced or metastatic cutaneous squamous cell carcinoma (cSCC) with 1 or more measurable lesions (greater than or equal to 1 cm).
* A history of either (Cohort 1) allogeneic hematopoietic stem cell transplant (alloHSCT) and ≥ 2 years or 730 days from day 0 of their HSCT with adequate bone marrow function (see Section 3.1.6) and off of all systemic immunosuppression (topical agents permitted) for at least 3 months prior to enrollment; sequelae of chronic graft versus host disease (GVHD) is permitted (i.e. chronic dry eyes, sclerodermatous skin changes, etc.) if the patient is not on systemic immunosuppression, or (Cohort 2) a renal transplant with a functioning allograft (at least 6 months from allograft transplant) as determined by estimated glomerular filtration (GFR) rate (CKD-EPI equation [40], Appendix A) ≥30 mL/min, baseline proteinuria lower than 0.5 g/day (spot urine protein-creatinine ratio), and off antiproliferative immunosuppressive medications.
* Age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix B).
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥ 2,200/mcL
  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 90,000/mcL
  * total bilirubin within normal institutional limits (except in cases where Gilbert syndrome is known or suspected, where total bilirubin should be < 3 mg/dL)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal
  * creatinine ≤ 1.5 × institutional upper limit of normal OR
  * estimated GFR ≥ 30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (CKD-EPI equation).
  * urine protein/creatinine ratio < 0.5 (equal to less than 500 mg of proteinuria per day)
* Ability to understand and the willingness to sign a written informed consent document.
* A prior history of acute GVHD that has resolved, or sequelae of chronic GVHD following allo-HSCT is permitted. Active acute GVHD patients are excluded.
* Women of childbearing potential (WOCBP) must agree to use at least 1 highly effective form of contraception (refer to Appendix C for examples). WOCBP should plan to use an adequate method to avoid pregnancy for up to 7 months (30 days plus the time required for cemiplimab to undergo five half-lives) after the last dose of investigational drug.

"Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche, who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy), who is not postmenopausal, who is sexually active with a male partner. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.

* Women of childbearing potential, as defined above, must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of cemiplimab.
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential as defined above, and azoospermic men) do not require contraception. See Appendix C for further guidance on contraception

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have unresolved toxicities from prior anti-cancer therapy more than 4 weeks earlier, defined as not resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 5.0), grade 0 or 1.
* Participants who are receiving any other investigational agents.
* For Cohort 1 allo-HSCT patients enrolling to the study, corticosteroid doses > 10 mg of prednisone daily or equivalent within 4 weeks of the first dose of PD-1 inhibitor are prohibited. For Cohort 2 renal transplant patients enrolling to the study, corticosteroid use is permitted if used as part of their immunosuppressive regimen for graft protection prior to enrollment.
* Existing significant autoimmune conditions. Patients with a history of Hashimoto thyroiditis who are stable on replacement hormone therapy are not excluded.
* Known human immunodeficiency virus carrier or a diagnosis of immunodeficiency. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
* Kidney transplant recipients with active acute rejection.
* Allergy to cemiplimab or any of its components.
* Any prior exposure to the phosphoinositide 3-kinase inhibitor idelalisib.
* Subject who has been treated with immunotherapy. This includes prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways (including chimeric antigen receptor [CAR] T cell therapies). Prior topical or intralesional immunotherapies (e.g. imiquimod, talimogene laherparepvec) are allowed.
* Subject with known and untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, baseline brain imaging is not required prior to enrollment in the study if patients are asymptomatic. Patients at least 4 weeks out from metastatic central nervous system (CNS) treatment are permitted to enroll, if they are asymptomatic, radiographically stable per the investigator, and on stable doses of anti-epileptic drugs (AEDs) and oral corticosteroids (for Cohort 1 only, the patient must be on 10 mg of prednisone daily equivalent dosing or less, see 3.2.2) at the time of enrollment.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as [http://medicine.iupui.edu/clinpharm/ddis/table.aspx]. Medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Known non-infectious pneumonitis or any history of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2025-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Hanna GJ, Dharanesswaran H, Giobbie-Hurder A, Harran JJ, Liao Z, Pai L, Tchekmedyian V, Ruiz ES, Waldman AH, Schmults CD, Riella LV, Lizotte P, Paweletz CP, Chandraker AK, Murakami N, Silk AW. Cemiplimab for Kidney Transplant Recipients With Advanced Cutaneous Squamous Cell Carcinoma. J Clin Oncol. 2024 Mar 20;42(9):1021-1030. doi: 10.1200/JCO.23.01498. Epub 2024 Jan 22. PMID 38252908
- [Derived] Bonilla M, Gudsoorkar P, Wanchoo R, Herrmann SM, Jhaveri KD. Onconephrology 2022: An Update. Kidney360. 2023 Feb 1;4(2):258-271. doi: 10.34067/KID.0001582022. Epub 2022 Dec 9. PMID 36821617
- [Derived] Paoluzzi L, Ow TJ. Safe Administration of Cemiplimab to a Kidney Transplant Patient with Locally Advanced Squamous Cell Carcinoma of the Scalp. Curr Oncol. 2021 Jan 19;28(1):574-580. doi: 10.3390/curroncol28010057. PMID 33477979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a phase I, single-arm, single-center, nonrandomized trial that enrolled patients at Dana-Farber Cancer Institute. The trial design originally included two parallel cohorts, one for allogeneic stem-cell transplant recipients and the other for patients with prior kidney transplantation. The stem-cell transplant cohort (Cohort 1) closed for slow accrual in November 2021 with no enrolled patients.
Groups:
- Cohort 1 Cemiplimab: Participants who received allogeneic hematopoietic stem cell transplant
  -- Cemiplimab: via IV, flat predetermined dosage every 21 days
  Cemiplimab: Cemiplimab: via IV, flat predetermined dosage every 21 days.
- Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone: Participants with a prior kidney transplant will receive
  * Cemiplimab via IV, flat predetermined dosage every 21 days
  * Everolimus or Sirolimus-least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  * Prednisone 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapering doses while receiving Cemiplimab
  Cemiplimab: Cemiplimab: via IV, flat predetermined dosage every 21 days.
  Everolimus: Everolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Sirolimus: Sirolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Prednisone: 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapered dosing while receiving Cemiplimab
Period: Overall Study
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Started | 0 | 12
Completed | 0 | 11
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: No patients were enrolled into Cohort 1.
Groups:
- Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone: Participants who received a kidney transplant will receive
  * Cemiplimab via IV, flat predetermined dosage every 21 days
  * Everolimus or Sirolimus-least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  * Prednisone 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapering doses while receiving Cemiplimab
  Cemiplimab: Cemiplimab: via IV, flat predetermined dosage every 21 days.
  Everolimus: Everolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Sirolimus: Sirolimus at least 7-10 days prior to receiving the first dose of cemiplimab (Cycle 1, Day 1) and then daily while receiving Cemiplimab
  Prednisone: 40 mg orally the day prior to the start of cemiplimab dosing (Cycle 1, Day 1) and then daily at tapered dosing while receiving Cemiplimab
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone | Total
Number analyzed (Participants) | 0 | 12 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] |  | 62.2 (12.6) | 62.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2
  Male |  | 10 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 11 | 11
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 11 | 11
  More than one race |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Years between initial diagnosis and enrollment [Median (Full Range); unit: Years] |  | 2.5 [0.2 to 4.6] | 2.5 [0.2 to 4.6]
Weeks between initial diagnosis and local or regional recurrence [Median (Full Range); unit: Weeks] |  | 70.4 [5.3 to 215.4] | 70.4 [5.3 to 215.4]
Site of recurrent disease [Count of Participants; unit: Participants]
  Regional |  | 8 | 8
  Local |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Rate of Renal Transplant Rejection (Cohort 2) or GVHD (Cohort 1).
Description: The proportions of patients who have observed GVHD in Cohort 1 or renal transplant rejection in Cohort 2.
  Participants will be evaluable for from the time of their first treatment.
Time Frame: First dose of study treatment up to 100 days
Population: No patients enrolled into Cohort 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Number analyzed (Participants) | 0 | 12
Percentage of participants |  | 0 [0 to 22.0]

2. Secondary Outcome: Progression-Free Survival
Description: Time from registration to the earlier of progression or death due to any cause. The follow-up of patients who neither progress nor die is censored at the date of last follow-up.
Time Frame: Duration of follow-up (up to 36 months)
Population: No patients enrolled into Cohort 1.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Number analyzed (Participants) | 0 | 12
Months |  | 22.5 [1.2 to 29.8]

3. Secondary Outcome: Overall Survival
Description: Time from registration to death due to any cause. Follow-up of patients who did not die will be censored at the date of last vital status.
Time Frame: Duration of follow-up (up to 36 months)
Population: No patients enrolled into Cohort 1.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Number analyzed (Participants) | 0 | 12
Months |  | 22.5 [2.9 to 29.8]

4. Secondary Outcome: Overall Response Rate
Description: The proportion of patients with best response of complete (CR) or partial (PR) response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 1 year
Population: Eleven of 12 patients had scans to assess RECIST response.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Number analyzed (Participants) | 0 | 11
Percentage of participants |  | 45.5 [20 to 73]

5. Secondary Outcome: Duration of Response
Description: Duration of response is estimated in the subset of patients with best response of complete or partial response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): at least 30% decrease in the sum of the longest diameter of target lesions. Duration of response is the time interval between dates of CR or PR and disease progression. The follow-up of patients who did not progress is censored at the date of the last follow-up scan.
Time Frame: Duration of follow-up (up to 36 months)
Population: Patients with best response of CR or PR per RECIST.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
Number analyzed (Participants) | 0 | 5
Months |  | 11.4 [4.9 to 29.7]

ADVERSE EVENTS:
Time Frame: All adverse events reported through study completion (up to 36 months).
Description: No patients enrolled into Cohort 1.
Arm/Group | Cohort 1 Cemiplimab | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone
All-Cause Mortality (participants affected / at risk) | 0/0 | 5/12
Serious Adverse Events (participants affected / at risk) | 0/0 | 9/12
Other Adverse Events (participants affected / at risk) | 0/0 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Cemiplimab (N=0) | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | NA | 1 (1)
Cardiac stent placement (Cardiac disorders) | NA | 1 (1)
Fever (General disorders) | NA | 1 (1)
Lung infection (Infections and infestations) | NA | 2 (2)
Skin infection (Infections and infestations) | NA | 1 (1)
Soft tissue infection (Infections and infestations) | NA | 1 (1)
Upper respiratory infection (Infections and infestations) | NA | 4 (4)
Creatinine increase (Investigations) | NA | 1 (1)
Acidosis (Metabolism and nutrition disorders) | NA | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | NA | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Hypotension (Vascular disorders) | NA | 1 (1)
Thromboembolic event (Vascular disorders) | NA | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Cemiplimab (N=0) | Cohort 2 Cemiplimab + Everolimus/Sirolimus + Prednisone (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (8)
Palpitations (Cardiac disorders) | NA | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | NA | 1 (1)
Hyperparathyroidism (Endocrine disorders) | NA | 1 (1)
Hyperthyroidism (Endocrine disorders) | NA | 2 (5)
Hypothyroidism (Endocrine disorders) | NA | 1 (2)
Eyelid function disorder (Eye disorders) | NA | 1 (1)
Watering eyes (Eye disorders) | NA | 1 (2)
Abdominal pain (Gastrointestinal disorders) | NA | 1 (1)
Constipation (Gastrointestinal disorders) | NA | 3 (5)
Diarrhea (Gastrointestinal disorders) | NA | 4 (10)
Dyspepsia (Gastrointestinal disorders) | NA | 2 (2)
Nausea (Gastrointestinal disorders) | NA | 2 (3)
Oral pain (Gastrointestinal disorders) | NA | 2 (2)
Vomiting (Gastrointestinal disorders) | NA | 1 (1)
Chills (General disorders) | NA | 1 (1)
Edema face (General disorders) | NA | 3 (3)
Edema limbs (General disorders) | NA | 6 (9)
Edema trunk (General disorders) | NA | 1 (1)
Facial pain (General disorders) | NA | 2 (2)
Fatigue (General disorders) | NA | 9 (19)
Fever (General disorders) | NA | 3 (4)
Flu like symptoms (General disorders) | NA | 1 (1)
Pain (General disorders) | NA | 1 (1)
Lung infection (Infections and infestations) | NA | 1 (1)
Nail infection (Infections and infestations) | NA | 1 (1)
Skin infection (Infections and infestations) | NA | 2 (4)
Thrush (Infections and infestations) | NA | 1 (1)
Urinary tract infection (Infections and infestations) | NA | 1 (2)
Wound infection (Infections and infestations) | NA | 2 (2)
Fall (Injury, poisoning and procedural complications) | NA | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | NA | 1 (1)
Alanine aminotransferase increased (Investigations) | NA | 3 (3)
Alkaline phosphatase increased (Investigations) | NA | 1 (2)
Aspartate aminotransferase increased (Investigations) | NA | 4 (5)
Cholesterol high (Investigations) | NA | 1 (1)
Creatinine increased (Investigations) | NA | 5 (15)
Platelet count decreased (Investigations) | NA | 2 (3)
Thyroid stimulating hormone increased (Investigations) | NA | 1 (1)
Anorexia (Metabolism and nutrition disorders) | NA | 2 (2)
Dehydration (Metabolism and nutrition disorders) | NA | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | NA | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | NA | 2 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | NA | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | NA | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | NA | 2 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | NA | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | NA | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | NA | 5 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | NA | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | NA | 2 (3)
Muscle cramp (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | NA | 1 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Dizziness (Nervous system disorders) | NA | 1 (1)
Headache (Nervous system disorders) | NA | 1 (2)
Paresthesia (Nervous system disorders) | NA | 1 (1)
Confusion (Psychiatric disorders) | NA | 1 (1)
Depression (Psychiatric disorders) | NA | 1 (1)
Insomnia (Psychiatric disorders) | NA | 4 (6)
Hematuria (Renal and urinary disorders) | NA | 1 (1)
Proteinuria (Renal and urinary disorders) | NA | 2 (7)
Urinary frequency (Renal and urinary disorders) | NA | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 3 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | NA | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | NA | 1 (1) — Crusting/dead debris on scalp
Flushing (Vascular disorders) | NA | 1 (1)
Hematoma (Vascular disorders) | NA | 1 (1)
Hypertension (Vascular disorders) | NA | 3 (4)
Lymphedema (Vascular disorders) | NA | 1 (1)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | NA | 2 (2)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | NA | 1 (1)

LIMITATIONS AND CAVEATS:
Limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04339062/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT04339062/SAP_001.pdf